CLINICAL TRIAL: NCT02962219
Title: A Pre-operative Personalised Exercise Programme to Improve Physical Fitness and Reduce Post-operative Cardiopulmonary Complications After Oesophagectomy in Patients With Oesophageal Adenocarcinoma: A Feasibility Randomised Controlled Trial
Brief Title: Exercise Prior to Oesophagectomy
Acronym: ExPO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of East Anglia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 206608
Record Dates: First submitted 2016-10-28; First posted 2016-11-11 (Estimated); Last update posted 2016-11-11 (Estimated); Status verified 2016-11

CONDITIONS: Postoperative Complications (Cardiopulmonary); Oesophageal Adenocarcinoma
Keywords: oesophagectomy
MeSH Terms: conditions — Postoperative Complications; Adenocarcinoma Of Esophagus

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Experimental): A pre-operative personalised exercise programme (my-PEP).
  Interventions: Behavioral: Pre-operative Exercise Programme (my-PEP)
- Control (Other): Standard care
  Interventions: Behavioral: Home Exercise Programme (HEP)

INTERVENTIONS:
Behavioral: Pre-operative Exercise Programme (my-PEP) — A pre-operative personalised exercise programme (my-PEP) consisting of: 1) actions to promote exercise, using behavioural change techniques (BCTs), 2) home inspiratory muscle training (IMT), 3) a home exercise programme (HEP) - which is also current standard care, 4) a 4 week hospital-supervised aerobic and muscle strengthening programme (Hos-PEP) .
  Arms: Intervention
Behavioral: Home Exercise Programme (HEP) — Written advice on exercise at home
  Arms: Control

SUMMARY:
The purpose of this feasibility study is to determine whether a structured exercise programme prior to oesophagectomy has: acceptable adherence, is safe, and improves physiological measures of physical fitness above standard care.

DETAILED DESCRIPTION:
The number of patients with oesophageal cancer is rising dramatically in the UK. Curative cancer surgery (oesophagectomy) is offered to around 40% of affected patients. However, oesophagectomy is a major operation with a high risk of complications. Around 1 in 3 patients will suffer such a complication after surgery, mostly due to heart or lung problems. Most complications are not due to the surgery itself, but related to the patient's physical fitness before their operation. Studies in other surgeries, but not oesophagectomy, have shown that complications may be reduced by improving a patient's physical fitness before their operation. The ExPO team has developed a pre-operative Personalised Exercise Programme (my-PEP), specifically for patients undergoing oesophagectomy. my-PEP has 4 main components: three are exercise modalities (aerobic exercise, breathing exercises and muscle strengthening); the fourth is where a participant's potential barriers to exercise are assessed and behavioural change techniques (BCTs) are suggested to improve exercise engagement in the trial. In total, 32 patients who are due to undergo oesophagectomy at the Norfolk and Norwich Hospital will be recruited and then randomly divided into 2 arms of 16 each. One arm will receive my-PEP in the standard 3-4 months prior to surgery, the other will receive standard care advice to exercise at home. The research objectives are to obtain feasibility data on whether my-PEP is acceptable, adhered to and safe, and whether it improves patient fitness above standard care. Follow up will be 90 days after surgery to obtain a preliminary imprecise estimate of whether my-PEP reduces complications. If the ExPO trial shows promise in these areas, this will inform and justify a future large multi-centre trial to definitively answer whether my-PEP can reduce complications after oesophagectomy. If so, my-PEP could potentially change and improve the pre-operative management of oesophageal cancer patients across the NHS.

ELIGIBILITY:
Inclusion Criteria:

* Patients with oesophageal adenocarcinoma (OAC) who are scheduled for neoadjuvant chemotherapy and subsequent oesophagectomy.
* Must have histological evidence of OAC
* Must be capable of giving informed consent and complying with trial procedures.

Exclusion Criteria:

* Patients with oesophageal squamous cell carcinoma.
* Patients with concomitant illness or disability that makes them unsuitable for an exercise programme, as determined by a clinician (e.g. severe musculoskeletal or neurological disease, unstable angina, severe aortic stenosis, uncontrolled dysrhythmias and uncompensated heart failure).
* WHO performance status 3 (capable of only limited self-care, confined to a bed or chair more that 50% of waking hours) or greater.
* Grade 5 (too breathless to leave the house, or breathless when undressing) on MRC dyspnoea scale.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2016-09; Primary Completion 2017-09 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate | 0 months
  The number of participants recruited from all eligible patients
Drop-out rate | 12 months
  Number of patients that drop-out from trial
Decline rate | 0 months
  Number of patients that decline to participate in the trial
Change in physical activity levels | 0 and 4 months
  Measured with International Physical Activity Questionnaire (IPAQ)
Change in attitudes to exercise | 0 and 4 months
  Measured with Determinates of Physical Activity Questionnaire (DPAQ)
Trial Adherence | 12 months
  Physical activity diary used to assess adherence
Adverse Events | 12 months
  The number of adverse events during the trial assessed using CTCAE
Change in physiological fitness | 0 and 4 months
  Assessed with maximal cardiopulmonary exercise test on a bicycle ergometer
Change in respiratory muscle strength | 0 and 4 months
  Assessed with mean inspiratory pressure testing in cmH20
Post-operative cardiopulmonary complications | 90-days post surgery
  Cardiopulmonary complication rates as per ECCG definition.
Post-operative non-cardiopulmonary complications | 90-days post surgery
  Inpatient, 30-day and 90-day non-cardiopulmonary complication rates as per ECCG definition.
Post-operative length of stay | 90-days post surgery
  Duration of post-operative stay in days
Post-operative mortality | 90-days post surgery
  Number of post-operative deaths
Change in Quality of Life | 0, 4, 7 months
  Assessed using QLQ C30 and OG25

CONTACTS AND LOCATIONS:
Locations (1):
- University of East Anglia, Norwich, Norfolk, United Kingdom

IPD SHARING:
Plan to Share IPD: No